CLINICAL TRIAL: NCT02686866
Title: Comparing Body Composition Measurements - Bioelectrical Impedance Analysis and Dual-energy X-ray Absorptiometry - in Chronic Heart Failure
Brief Title: Body Composition Measurements in Chronic Heart Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hungarian Institute of Cardiology (Other Government)
Responsible Party: Principal Investigator, ANDREKA PETER, MD, PhD, FESC, Hungarian Institute of Cardiology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 101568/2015/OTIG
Record Dates: First submitted 2016-02-02; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Cachexia; Sarcopenia; Body Composition
MeSH Terms: conditions — Cachexia; Sarcopenia | interventions — Absorptiometry, Photon; Hand Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Body composition measurement (Experimental): All patients will undergo body composition measurement with dual-energy X-ray absorptiometry and bioelectrical impedance analysis methods. Hand grip strength will also be performed.
  Interventions: Device: bioelectrical impedance analysis (Bodystat, Quadscan 4000); Device: dual-energy X-ray absorptiometry (Hologic, Delphi QDR); Device: hand grip strength

INTERVENTIONS:
Device: bioelectrical impedance analysis (Bodystat, Quadscan 4000)
Device: dual-energy X-ray absorptiometry (Hologic, Delphi QDR)
Device: hand grip strength

SUMMARY:
Feeding optimization and nutritional assessment in patients with severe heart failure are challenging. The prevalence of cardiac cachexia may be underestimated by simple measurements of body weight and body mass index because many patients show relative reductions in muscle mass despite being of normal overall weight. Body composition measurement can be essential in chronic heart failure (CHF) patients to estimate sarcopenia. Chronic heart failure patients with cardiac cachexia have a mortality two to three times higher than noncachectic patients. Bedside body composition measurements can reveal developing cardiac cachexia hence can be useful in prevention.

DETAILED DESCRIPTION:
Feeding optimization and nutritional assessment in patients with severe heart failure are challenging. The reasons are rather complex and many questions have not been answered yet. Unfortunately, no clear and definitive guidelines are available from the big Nutritional Societies - The European Society for Clinical Nutrition and Metabolism (ESPEN), American Society for Parenteral and Enteral Nutrition (ASPEN), British Association for Parenteral and Enteral Nutrition (BAPEN), Society of Critical Care Medicine (SCCM), Canadian Clinical Care Guidelines. However, there are more and more heated debates in Nutritional Conferences and the need of "Heart Failure feeding-guidelines" is urged. Though local and international comprehensive proposals are highly demanded unfortunately these suggestions are still missing. As we mentioned above there are lots of reasons why this nutritional insufficiency persists. Probably one of these reasons is the "splitting" of medical professions hence creating a proper guideline entail many problems and reveal some unsought difficulties such as lack of knowledge.

The nutrition (esp. TPN) primarily is carried out by anaesthetists and in a less extent manner by gastroenterologists. Feeding performed by surgeons, internists, paediatricians etc. is minimal. Cardiologists can play an important role in the field of nutrition. Cardiac patients are losing their weights very easily and their cardiac cachexia is usually not perceived by most of cardiologists. The best conceivable compensation of heart failure is a prerequisite of "nutritional appropriateness" and in most severe cases this compensation is done by cardiologists. Without this compensation and consequently insufficient cardiac output, this "refeeding" seems to be impossible. Cardia cachexia is an absolute contraindication of Heart Transplantation (HTX) and Ventricular Assist Device/Total Artificial Heart (VAD/TAH) implantation. These patients are usually younger than 65 year-of-age, the expected quality of life (QoL) with a transplanted heart is good and according to the international data the rate of survival is acceptable. Moreover, it is a well known phenomenon that the prevention of cardiac cachexia is much easier than its treatment. Sadly, the use of known nutritional scoring systems - Malnutrition Universal Screening Tool (MUST), Short Nutritional Assessment Questionnaire (SNAQ), Nutritional Risk screening (NRS2002), Malnutrition Screening Tool (MST), Subjective Global Assessment (SGA), Mini Nutritional Assessment (MNA) - which work well in other situations, are of limited value or might not be used at all in this patient group. We must emphasize the fact that increasing number of patients suffering in end-stage heart disease (ESHD) can be expected and further specialization within cardiology makes this problem more pronounced. Without this proper compensation appropriate nutrition is often impossible as well as cardiac compensation can be unsuccessful without proper feeding.

The existing recommendations and traditions in gastroenterology and surgery are different hence it seems to be sensible that the formentioned facts may contribute to the lack of proper guidelines. We believe that the elimination of cardiac cachexia is feasible only with special care and in suitable units. In 2014 our ICU patients, who had not previously been eligible for HTX because of their cachexia, were treated according to our "protocol" and all of them reached the minimum desired weight and were transplanted. The postoperative care and recuperation was similar to those who had not been suffered from cachexia before. These results were also similar we found in the literature. According to our experiences cardiac cachexia seems to be manageable. In case of proper nutrition, international cost-benefit analyses showed positive results regarding patients' recovery: less infections and severe sepsis, decreasing number of in-hospital stays, better wound healing and less ventilatory and ICU days.

Summing up we would like to draw the attention for an unsolved problem which exists not only in Hungary but all over the world. The solution of this problem is urgent but seems possible. We think for overcoming this severe condition we have to change our system, we need new guidelines, we need education and we need further research.

The definition of cardiac cachexia is weight loss of 6% or more in at least 6 months. The incidence in CHF patients with NYHA class III/IV is approximately 10% per year. Chronic heart failure patients with cardiac cachexia have a mortality two to three times higher than noncachectic patients. The prevalence of cardiac cachexia may be underestimated by simple measurements of body weight and body mass index because many patients show relative reductions in muscle mass despite being of normal overall weight. Body composition measurement can be essential in chronic heart failure patients to estimate sarcopenia. These methods can determine the different components of the whole body weight. To estimate sarcopenia it is essential to measure fat-free mass (FFM). According to literature dual energy X-ray absorptiometry (DXA) is the gold standard procedure to determine body composition and FFM. The use of DXA is limited in chronic heart failure patients due to low availability and relatively high cost. Bioelectrical impedance analysis (BIA) is a non-invasive, relatively low cost, bedside body composition measurement method. With no radiation exposure it can be repeated multiple times.

Hypothesis:

The BIA method is already validated in healthy patients and in different disease groups. We suppose that it can be used and reliable data can be obtained in chronic heart failure patient population.

Objectives and aims:

Bioelectrical impedance analysis is not approved in extreme body mass index and body fluid ranges. These conditions however may present in chronic heart failure patients. Thus it is essential to validate BIA to the gold standard DXA method which is our primary aim. Patients admitted to Gottsegen György Hungarian Institute of Cardiology with acute decompensation of chronic heart failure will be enrolled in this prospective study. Enrolled participants will undergo body composition measurements with dual-energy X-ray absorptiometry (Hologic, Delphi QDR) and bioelectrical impedance analysis (Bodystat, Quadscan 4000) methods. The main measured parameters - body weight, total body water, fat mass, fat-free mass (lean weight), extracellular mass, body cell mass, resistance, reactance, phase angle, basal metabolic rate - will be registered in database. Statistical analysis of data acquired by the different methods will be performed to validate BIA.

Primary aim:

1. Verify that bioelectrical impedance analysis can be safely performed in chronic heart failure patients.
2. Compare body composition values measured with BIA and DXA. Validate the use of BIA in chronic heart failure patient population.

Secondary aim:

To examine if there is a relationship between sarcopenia or any other altered body composition value and other parameters of chronic heart failure (NYHA functional class, biomarkers, echocardiographic values, hand grip test).

Expected results:

Body composition values measured by bioelectric impedance analysis are correlating with DXA values. These results validate the use of BIA in chronic heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure (NYHA III-IV)
* Hospitalization for acute decompensation
* Willing to participate

Exclusion Criteria:

* Unstable hemodynamic status
* Iv. inotropic, vasopressor support
* Severe orthopnea
* Pacemaker, implantable cardioverter-defibrillator (ICD), cardiac resynchronization therapy (CRT)
* High fever
* Contrast agent administration within 1 week
* Females with childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Compare total body water (TBW) measured with BIA and DXA. | 6 month
Compare fat mass (FM) measured with BIA and DXA. | 6 month
Compare fat-free mass (FFM) measured with BIA and DXA. | 6 month
Compare extracellular mass (ECM) measured with BIA and DXA. | 6 month
Compare body cell mass (BCM) measured with BIA and DXA. | 6 month

SECONDARY OUTCOMES:
Evaluate adverse events that are related to study procedure. | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Peter Andreka, MD, PhD, Principal Investigator — Hungarian Institute of Cardiology
Locations (1):
- Hungarian Institute of Cardiology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided